CLINICAL TRIAL: NCT01247142
Title: Evaluation of Exhaled Breath Condensate in the Diagnosis of Invasive Pulmonary Aspergillosis
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Edith Vermeulen, PhD fellow, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S52756
Record Dates: First submitted 2010-11-23; First posted 2010-11-24 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Invasive Pulmonary Aspergillosis
Keywords: invasive pulmonary aspergillosis; exhaled breath condensate
MeSH Terms: conditions — Invasive Pulmonary Aspergillosis

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — exhaled breath condensate
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Invasive pulmonary aspergillosis (IPA): Patients with proven or probable invasive pulmonary aspergillosis (IPA) (EORTC/MSG criteria) or putative IPA (Blot et al. Am J Respir Crit Care Med 2012)
- Controls: Patients without signs of infection.

SUMMARY:
The purpose of this study is to evaluate the diagnostic potential of biomarkers for invasive pulmonary aspergillosis in exhaled breath condensate.

DETAILED DESCRIPTION:
Invasive pulmonary aspergillosis (IPA) is a life-threatening infection in immunocompromised patients. The poor prognosis of the disease is partly attributed to difficulties encountered with the diagnosis of this infection. Invasive sampling procedures are often precluded in these patients. In addition, conventional diagnostic techniques lack sensitivity. Recently there has been increasing interest in the investigation of the lungs by noninvasive means including measurement of biomarkers in exhaled breath (e.g. NO) and those found in the cooled and condensed exhalate,termed EBC. It has been demonstrated that a measurable fraction of the EBC in healthy subjects is derived from aerosolized airway lining fluid. The presence of biomarkers for IPA will be investigated in EBC of patients with IPA, compared to controls.

ELIGIBILITY:
Inclusion Criteria:

* hospitalisation in the hematology or intensive care department
* age > 16 years
* informed consent
* proven or probable IPA (EORTC/ MSG criteria)
* galactomannan positivity in BAL or serum

Exclusion Criteria:

* age < 16 years

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized adult patients of the department of Hematology or Intensive Care Unit, University Hospital, Leuven, Belgium
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2011-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The identification of biomarkers for invasive pulmonary aspergillosis (IPA) in exhaled breath condensate (EBC) | 15 months

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium